CLINICAL TRIAL: NCT04814901
Title: Patient Satisfaction After Using Reverse Flow Based Facial Artery Musculomucosal Flap (FAMM) Versus Palatal Pedicled Flap for Closure of Recurrent Small and Medium Sized Oronasal Fistula. A Randomized Clinical Trial.
Brief Title: Using Reverse Flow Based Flap VS Palatal Pedicled Flap for Closure of Recurrent Small & Medium Sized Oronasal Fistula.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Doaa Jawad Roomi (Other)
Responsible Party: Sponsor-Investigator, Doaa Jawad Roomi, Principal Investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OMFS 3-3-8
Record Dates: First submitted 2021-03-11; First posted 2021-03-24 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: 2 arms parallel group of patients will be assigned to this trial: The trial will be in superiority in an allocation of 1:1 ratio.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Surgical closure of patients with recurrent small to medium sized oronasal fistulae using FAMM and assessment of success regarding patient satisfaction and healing and absence of complications such as venous congestion, dehiscence, facial nerve injury and infection.
  Interventions: Procedure: Curing small and medium sized oronasal fistula
- Comparator group (Active Comparator): Surgical closure of patients with recurrent small to medium sized oronasal fistulae and its effect on patient's satisfaction and healing and absence of complications such as venous congestion, dehiscence, facial nerve injury and infection
  Interventions: Procedure: Curing small and medium sized oronasal fistula

INTERVENTIONS:
Procedure: Curing small and medium sized oronasal fistula — * Flap will be marked medial to the duct, which limits posterior extent of flap. Anterior flap marking starts 1cm posterior to oral commissure.
  * Width of flap was kept to about 2-2.5cm.
  * An initial incision will be made 1cm posterior to oral commissure.
  * Incision will be deepened through buccal mucosa, submucosa, & underlying muscles into layer of buccal fat.
  * Flap will be dissected in a retrograde or antegrade manner depending on fistula site, maintaining vessels in a central position in the flap.
  * Once completely raised, flap inserted & sutured in place while donor site be closed primarily with 4-0 polyglactin (Vicryl) interrupted sutures.
  * Patient's comparator group will be treated by raising a palatal pedicled flap.
  * Flap will be outlined extending from palatal mucosa against permanent 2nd molar till permanent canine anteriorly.
  * It is rotated towards oronasal fistula & secured in place using 4 -0 Vicryl interrupted sutures.

SUMMARY:
Research question:

What are the outcomes of using the Facial artery Musculomucosal (FAMM) Flap to close recurrent small and medium sized oronasal fistulae based on reverse flow on patient's satisfaction versus using the Palatal Pedicled flap?

Statement of the problem:

To determine whether the using the Facial artery Musculomucosal (FAMM) Flap to close recurrent small and medium sized oronasal fistulae which are difficult to manage could meet the patients satisfaction regarding both success and function versus using palatal pedicled flap

DETAILED DESCRIPTION:
Oronasal fistulae (particularly those of the anterior palate) are often difficult to close because the buccal cavity is narrow and the palatal mucosa is not extensible.

Historically, skin flaps (forehead or nasolabial skin flaps) were first used to close such defects. but they leave a conspicuous scar. Mucosal flaps, which were empirically harvested from the cheek mucosa have also been used occasionally, but unpredictable results discouraged further attempts. A more accurate description of the vascularization of the buccal mucosal has allowed the design of axial-pattern flaps. The buccinator musculomucosal flap was first introduced as an island flap supported by the facial pedicle, and was then used successfully as an axial pattern flap that was vascularized by the buccal artery according to Bozola et al. or the facial artery according to Carstens et al.

The FAMM (facial artery musculomucosal) flap was introduced by Pribaz et al. in 1992 and its main advantage is its long rotational arc that allows closure of defects of the anterior palate that were formerly a reconstructive challenge. Pribaz et al. gave an accurate description of the dissection of the flap, but variations in the course of the facial artery sometimes preclude its use. Previous studies involving FAMM flap were applied to oronasal fistula repair either recurrent or as first attempt were described in repair of alveolar clefts, anterior palatal fistulae and in recurrent fistulae after palatoplasty in cleft patients either superior or inferior pediceled flap. In cases of hypovascular bed, it increases the chances for failure of other techniques of closure. The palatal pedilced flap was reported in the literature as one of the regional flaps for closure of oronasal fistulae. The previous studies included case series, with no any randomized clinical trial.

This study compares using FAMM flap versus Palatal Pedicled flap in a randomized clinical trial in closure of recurrent oronasal fistulae.

Aim of the study To evaluate the effect of using FAMM for closure of recurrent small and medium sized oronasal fistula on patient's satisfaction versus using the palatal pedicled flap.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent small and medium sized oronasal fistula failed after several attempts closure, up to 10 mm regardless of number of recurrence and position of the fistula.
* Age group : from 18 to 60 years old.
* No sex predilection.
* Patients with no contraindications to surgical intervention.
* Patients accepting consent for extracting one teeth in the surgical field if needed.
* Patients proved with Doppler study with a patent facial artery course.

Exclusion Criteria:

* Patients with systemic condition counteracting with the surgical procedure.
* Patients who underwent a previously ipsilateral cheek flap except for midline fistulae.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
questionnaire | 3 months
  Meet the patients satisfaction regarding both success and function after closure of recurrent small and medium sized oronasal fistula using the Facial artery Musculomucosal (FAMM) Flap

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith DM, Vecchione L, Jiang S, Ford M, Deleyiannis FW, Haralam MA, Naran S, Worrall CI, Dudas JR, Afifi AM, Marazita ML, Losee JE. The Pittsburgh Fistula Classification System: a standardized scheme for the description of palatal fistulas. Cleft Palate Craniofac J. 2007 Nov;44(6):590-4. doi: 10.1597/06-204.1. PMID 18177198
- [Background] Xiong B, Zhao M, Cheng T, Gao P. [Analysis of 5459 cleft lip and palate cases]. Zhonghua Zheng Xing Wai Ke Za Zhi. 2002 Sep;18(5):294-6. Chinese. PMID 12471822
- [Background] Wang HT, Li F. [Clinical study on fistula incidence of early cleft palate repair]. Zhonghua Zheng Xing Wai Ke Za Zhi. 2003 May;19(3):192-4. Chinese. PMID 12958822
- [Background] Richardson S, Agni NA. Palatal fistulae: a comprehensive classification and difficulty index. J Maxillofac Oral Surg. 2014 Sep;13(3):305-9. doi: 10.1007/s12663-013-0535-2. Epub 2013 May 26. PMID 25018605
- [Background] Cohen SR, Kalinowski J, LaRossa D, Randall P. Cleft palate fistulas: a multivariate statistical analysis of prevalence, etiology, and surgical management. Plast Reconstr Surg. 1991 Jun;87(6):1041-7. PMID 2034725
- [Background] Dupoirieux L, Plane L, Gard C, Penneau M. Anatomical basis and results of the facial artery musculomucosal flap for oral reconstruction. Br J Oral Maxillofac Surg. 1999 Feb;37(1):25-8. doi: 10.1054/bjom.1998.0301. PMID 10203218
- [Background] Jackson IT. Closure of secondary palatal fistulae with intra-oral tissue and bone grafting. Br J Plast Surg. 1972 Apr;25(2):93-105. doi: 10.1016/s0007-1226(72)80028-6. No abstract available. PMID 4554003
- [Background] Rayner CR. Oral mucosal flaps in midfacial reconstruction. Br J Plast Surg. 1984 Jan;37(1):43-7. doi: 10.1016/0007-1226(84)90039-0. PMID 6692059
- [Background] Sasaki TM, Taylor L, Martin L, Baker HW, McConnell DB, Vetto RM. Correction of cervical esophageal stricture using an axial island cheek flap. Head Neck Surg. 1983 Sep-Oct;6(1):596-9. doi: 10.1002/hed.2890060110. PMID 6629796
- [Background] Bozola AR, Gasques JA, Carriquiry CE, Cardoso de Oliveira M. The buccinator musculomucosal flap: anatomic study and clinical application. Plast Reconstr Surg. 1989 Aug;84(2):250-7. doi: 10.1097/00006534-198908000-00010. PMID 2748738
- [Background] Pribaz J, Stephens W, Crespo L, Gifford G. A new intraoral flap: facial artery musculomucosal (FAMM) flap. Plast Reconstr Surg. 1992 Sep;90(3):421-9. doi: 10.1097/00006534-199209000-00009. PMID 1513887
- [Background] Ariffuddin I, Arman Zaharil MS, Wan Azman WS, Ahmad Sukari H. The use of facial artery musculomucosal (FAMM) readvancement flap in closure of recurrent oronasal fistula. Med J Malaysia. 2018 Apr;73(2):112-113. PMID 29703876
- [Background] Yilmaz T, Suslu AE, Gursel B. Treatment of oroantral fistula:experience with 27 cases. Am J Otolaryngol. 2003 Jul-Aug;24(4):221-3. doi: 10.1016/s0196-0709(03)00027-9. PMID 12884211
- [Background] Shetty R, Lamba S, Gupta AK. Role of facial artery musculomucosal flap in large and recurrent palatal fistulae. Cleft Palate Craniofac J. 2013 Nov;50(6):730-3. doi: 10.1597/12-115. Epub 2013 Feb 18. PMID 23418920
- [Background] Ashtiani AK, Emami SA, Rasti M. Closure of complicated palatal fistula with facial artery musculomucosal flap. Plast Reconstr Surg. 2005 Aug;116(2):381-6; discussion 387-8. doi: 10.1097/01.prs.0000142475.63276.87. PMID 16079659
- [Background] Sohail M, Bashir MM, Khan FA, Ashraf N. Comparison of Clinical Outcome of Facial Artery Myomucosal Flap and Tongue Flap for Closure of Large Anterior Palatal Fistulas. J Craniofac Surg. 2016 Sep;27(6):1465-8. doi: 10.1097/SCS.0000000000002773. PMID 27526234
- [Background] Lahiri A, Richard B. Superiorly based facial artery musculomucosal flap for large anterior palatal fistulae in clefts. Cleft Palate Craniofac J. 2007 Sep;44(5):523-7. doi: 10.1597/06-164.1. PMID 17760492
- [Background] Rauso R, Tartaro G, Califano L, Rugge L, Chirico F, Colella G. Pedicled palatal flap for surgical repair of oro-nasal fistula. J Biol Regul Homeost Agents. 2018 Nov-Dec;32(6):1565-1567. PMID 30574765
- See also: Myomucosal island flap of the buccinator Muscle: An anatomical study — https://www.researchgate.net/publication/344719685_Myomucosal_island_flap_of_the_buccinator_Muscle_An_anatomical_study